CLINICAL TRIAL: NCT02146677
Title: Effect of Osteopathic Manipulative Treatment on Pain in Preterms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: European Institute for Evidence Based Osteopathic Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEO-Pa 1
Record Dates: First submitted 2014-05-20; First posted 2014-05-26 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Prematurity
Keywords: prematurity; newborns; pain; cost
MeSH Terms: conditions — Premature Birth; Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sham (Other): newborns will be osteopathically evaluated and softly touched
  Interventions: Other: Sham therapy; Other: Usual care
- Usual care (Other): newborns will be undergone usual routine neonatology care
  Interventions: Other: Usual care
- OMT (Other): newborns will receive osteopathic evaluation and treatment according to international guidelines. Osteopathic treatment use will be indirect techniques.
  Interventions: Other: Osteopathic manipulative treatment; Other: Usual care

INTERVENTIONS:
Other: Osteopathic manipulative treatment
  Arms: OMT
Other: Sham therapy
  Arms: Sham
Other: Usual care

SUMMARY:
Osteopathic manipulative treatment (OMT) has been used to treat term and preterm newborns. Recent studies demonstrated the effectiveness of OMT in reducing length of stay and costs (Cerritelli, 2013) as well as the likelihood of gastrointestinal episodes (Pizzolorusso 2011). Moreover it was reported the absence of adverse events and side effects considering the approach safe (Cerritelli 2013, 2014).

OMT was extensively used to treat, prevent and manage pain symptoms. Numerous research was published addressing acute and chronic pain in different medical conditions. However, no trials were carried out on pain in newborns. The aim of the present clinical trial is to explore the effectiveness of OMT in reducing pain in a sample of preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants
* written informed consent by parents or legal guardians
* preterms born in the same hospital

Exclusion Criteria:

* Gestational age > 37 weeks
* genetic disorders
* congenital disorders
* cardiovascular abnormalities
* proven or suspected necrotized enterocolitis with or without gastrointestinal perforation
* proven or suspected abdominal obstruction
* pre/post surgery patients
* pneumoperitoneum
* atelectasis
* Newborn from an HIV seropositive/drug addicted mother
* respiratory disorders
* transferred to/from other hospital
* admitted for preterminal comfort care (defined as neither intubation nor cardio-respiratory resuscitation)

Ages: 26 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
changes from baseline in pain using Premature Infant Pain Profile (PIPP) | baseline and end of hospitalization, average length of hospitalization expected 4 weeks

SECONDARY OUTCOMES:
Number of days of length of stay | participants will be followed for the duration of hospital stay, an expected average of 4 weeks

OTHER OUTCOMES:
Neonatal intensive care unit cost | participants will be followed for the duration of hospital stay, an expected average of 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Pescara Civil Hospital, Pescara, PE, Italy

REFERENCES:
- [Derived] Cerritelli F, Cicchitti L, Martelli M, Barlafante G, Renzetti C, Pizzolorusso G, Lupacchini M, D'Orazio M, Marinelli B, Cozzolino V, Fusilli P, D'Incecco C. Osteopathic manipulative treatment and pain in preterms: study protocol for a randomised controlled trial. Trials. 2015 Mar 8;16:84. doi: 10.1186/s13063-015-0615-3. PMID 25872943